CLINICAL TRIAL: NCT07012772
Title: COMBO Endoscopy Oropharyngeal Airway in Sedated Endoscopic Retrograde Cholangiopancreatography for Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025B0632
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Choledocholithiasis With Cholecystitis With Obstruction; Obstructive Jaundice; Pancreatitis; Cholelithiasis
Keywords: respiratory depression; The COMBO Endoscopy Oropharyngeal Airway; Hypoxia; Sedation; ERCP
MeSH Terms: conditions — Jaundice, Obstructive; Pancreatitis; Cholelithiasis; Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The COMBO Endoscopy Oropharyngeal Airway Group (Experimental): In this group, patients use the COMBO Endoscopy Oropharyngeal Airway for oxygenation.
  Interventions: Device: The COMBO Endoscopy Oropharyngeal Airway

INTERVENTIONS:
Device: The COMBO Endoscopy Oropharyngeal Airway — Using the COMBO Endoscopy Oropharyngeal Airway for oxygenation.

SUMMARY:
Hypoxia represents the prevailing adverse occurrence during the sedation of patients undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) with propofol. A recent innovation in this domain is the COMBO Endoscopy Oropharyngeal Airway-a multifaceted device that encompasses capnography monitoring, bite block , oxygenation support, and oropharyngeal airway management. This device has been purposefully designed to cater to the unique requirements of endoscopic procedures. The principal objective of this study is to assess the efficacy of the COMBO Endoscopy Oropharyngeal Airway in reducing the incidence of hypoxia in patients undergoing ERCP under sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years；
* The ASA classification ranges from I to III.
* Patients have signed the informed consent form.
* Patients scheduled to undergo sedated ERCP examination;
* The estimated duration of the procedure does not exceed 45 minutes.

Exclusion Criteria:

1. Patients with coagulation disorders, tendency for oral/nasal bleeding, mucosal injury/occupying lesions, or difficult oropharyngeal airway insertion making airway management unfeasible;
2. Severe cardiac dysfunction (<4 METs);
3. Severe renal insufficiency (requiring preoperative dialysis);
4. Child-Pugh class C;
5. Diagnosed chronic obstructive pulmonary disease (COPD) or other acute/chronic pulmonary diseases requiring long-term/intermittent oxygen therapy;
6. Increased intracranial pressure;
7. Upper respiratory tract infections (oral/nasal/pharyngeal);
8. Fever (core temperature >37.5°C);
9. Confirmed pregnancy or current breastfeeding;
10. Allergy to sedatives (e.g., propofol) or medical adhesives;
11. Emergency procedures;
12. Multiple trauma injuries;
13. Peripheral oxygen saturation (SpO2) levels below 95% while breathing room air preoperatively;
14. BMI <18.5 or >30 kg/m²;
15. Current participation in other clinical trials;
16. Other conditions deemed ineligible by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  75% ≤ SpO2 < 90% for <60 s

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90% ≤ SpO2 < 95%
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - he First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided